CLINICAL TRIAL: NCT03236922
Title: Pubococcygeus Versus Rectus Sheath Sling for Goh Class 3 and 4 Vesico-vaginal Fistulas: a Randomized Controlled Trial
Brief Title: Autologous Slings With Vesico-Vaginal Fistula Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jeffrey Wilkinson, Professor of Obstetrics and Gynecology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-38672
Record Dates: First submitted 2016-08-21; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Vesicovaginal Fistula
Keywords: obstetric fistula, anti-incontinence techniques
MeSH Terms: conditions — Vesicovaginal Fistula

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pubococcygeus Sling (Active Comparator): This is one anti-incontinence technique commonly used at the time of fistula surgery.
  Interventions: Procedure: Pubococcygeus sling
- Rectus Fascia Sling (Active Comparator): This is another anti-incontinence technique used at the time of fistula surgery, however, less commonly than the pubococcygeus.
  Interventions: Procedure: Rectus fascia sling

INTERVENTIONS:
Procedure: Pubococcygeus sling — The pubococcygeus muscles is dissected from the vaginal side walls and approximated at the midline just below the urethra.
  Other Names: pubococcygeal sling; pubococcygeus graft
  Arms: Pubococcygeus Sling
Procedure: Rectus fascia sling — Rectus fascia is dissected out cephalad to the pubic symphysis and tunneled beneath the urethra.
  Other Names: rectus fascia graft
  Arms: Rectus Fascia Sling

SUMMARY:
It is clear from multiple accounts in the literature that patients with a vesico-vaginal fistula (VVF) involving the bladder neck and/or proximal urethra have a high likelihood of residual incontinence. Performing subsequent surgeries after the initial VVF repair risks additional complications. Therefore, placement of an autologous sling at the time of initial VVF repair would not only assist in covering the fistula, but would also imitate the physiologic support that would theoretically improve urethral function. A rectus fascia sling would most naturally provide this support and warrants testing against the success of the PC sling.

Using the Goh scoring criteria, Goh class 3 and 4 VVF's are the type most involving the urethra. Therefore, this group of patients is the target population for this study. As there is currently no standard of care for repairing large urethral defects, this procedural technique combined with otherwise standardized fistula repair would not introduce any foreseeable harm to patients.

ELIGIBILITY:
Inclusion Criteria:

* Women with vesico-vaginal fistulas classified as Goh 3 or 4 at the time of surgery
* Patients who have consented for an autologous sling
* Patients who have not previously undergone repair attempt

Exclusion Criteria:

* Patients who require an abdominal approach to the VVF repair
* Patients found at surgery not to have a Goh 3 or 4 class VVF
* Patients requiring a complete urethral reconstruction
* Patients who have undergone previous attempt at repair
* Patients who require an alternative tissue grafting other than the rectus fascia or pubbococcygeus decided by the surgeon at the time of surgery

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-06; Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Long-term Continence Status | Six months after surgery
  Residual stress incontinence is commonly experienced by this patient population, therefore a dye test to ensure the fistula is still closed and a cough test to determine any incontinence will be performed.

SECONDARY OUTCOMES:
Vesico-vaginal fistula repaired | One month after surgery
  To ensure the VVF is still closed and was not compromised due to the sling

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pope, MD, MPH, Study Director — Baylor College of Medicine
Locations (1):
- Fistula Care Center, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Yes
No.

REFERENCES:
- [Background] Ascher-Walsh CJ, Capes TL, Lo Y, Idrissa A, Wilkinson J, Echols K, Crawford B, Genadry R. Sling procedures after repair of obstetric vesicovaginal fistula in Niamey, Niger. Int Urogynecol J. 2010 Nov;21(11):1385-90. doi: 10.1007/s00192-010-1202-5. Epub 2010 Jun 17. PMID 20556597
- [Result] Browning A. Risk factors for developing residual urinary incontinence after obstetric fistula repair. BJOG. 2006 Apr;113(4):482-5. doi: 10.1111/j.1471-0528.2006.00875.x. Epub 2006 Feb 20. PMID 16489933
- [Result] Browning A. Prevention of residual urinary incontinence following successful repair of obstetric vesico-vaginal fistula using a fibro-muscular sling. BJOG. 2004 Apr;111(4):357-61. doi: 10.1111/j.1471-0528.2004.00080.x. PMID 15008773
- [Result] Carey MP, Goh JT, Fynes MM, Murray CJ. Stress urinary incontinence after delayed primary closure of genitourinary fistula: a technique for surgical management. Am J Obstet Gynecol. 2002 May;186(5):948-53. doi: 10.1067/mob.2002.122247. PMID 12015520
- [Derived] Pope R, Browning A, Chipungu E, George JOM, Tamimu M, Wilkinson J. Prophylactic Autologous Slings at the Time of Obstetric Fistula Repair: A Randomized Clinical Trial. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):78-84. doi: 10.1097/SPV.0000000000000745. PMID 31145227